CLINICAL TRIAL: NCT01134900
Title: Achieving Medication Safety During Acute Kidney Injury: The Impact of Clinical Decision Support and Real-Time Pharmacy Surveillance
Brief Title: Achieving Medication Safety During Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Allison McCoy, Principle Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 081002; R01LM009965 (NIH)
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Failure, Acute
Keywords: Medication Errors; Adverse Drug Events; Decision Support Systems, Clinical
MeSH Terms: conditions — Acute Kidney Injury; Drug-Related Side Effects and Adverse Reactions | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dashboard (Experimental): Patients appear on dashboard and are eligible for pharmacy intervention in addition to existing clinical decision support interventions.
  Interventions: Other: Pharmacy Dashboard Review and Intervention
- Control (No Intervention): Patients do not appear on dashboard for pharmacy intervention, but only receive existing clinical decision support interventions.

INTERVENTIONS:
Other: Pharmacy Dashboard Review and Intervention — Clinical pharmacist reviews patients on dashboard and makes intervention with providing team when necessary.
  Arms: Dashboard

SUMMARY:
The utilization of clinical decision support (CDS) is increasing among healthcare facilities which have implemented computerized physician order entry or electronic medical records. Formal prospective evaluation of CDS implementations occurs rarely, and misuse or flaws in system design are often unrecognized. Retrospective review can identify failures but is too late to make critical corrections or initiate redesign efforts. A real-time surveillance dashboard for high-alert medications integrates externalized CDS interactions with relevant medication ordering, administration, and therapeutic monitoring data. The surveillance view of the dashboard displays all currently admitted, eligible patients and provides brief demographics with triggering order, laboratory, and CDS failure data to allow prioritization of high-risk scenarios. The patient detail view displays a detailed timeline of orders, order administrations, laboratory values, and CDS interactions for an individual patient and allows users to understand provider actions and patient condition changes occurring in conjunction with CDS failures. Clinical pharmacists' use of the dashboard for patient monitoring and intervention aims to increase the rate and timeliness of intercepted medication errors compared to CPOE-based CDS in the setting of acute kidney injury, which affects patients at various points across all hospital units and services and has numerous opportunities for intervention.

ELIGIBILITY:
Inclusion Criteria:

* 0.5 mg/dl increase or decrease in serum creatinine within 48 hours
* Active, recurring order for targeted renally cleared or nephrotoxic medication

Exclusion Criteria:

* Chronic dialysis
* Transplant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison B McCoy, PhD, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth); Josh F Peterson, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] McCoy AB, Peterson JF, Gadd CS, Danciu I, Waitman LR. A system to improve medication safety in the setting of acute kidney injury: initial provider response. AMIA Annu Symp Proc. 2008 Nov 6:1051. PMID 18999252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We performed a randomized, controlled trial during June 1, 2010 through August 31, 2010 at a large academic, tertiary care facility. We included all admitted adult patients who experienced a 0.5 mg/dl change in serum creatinine over 48 hours following an active, recurring order for one or more targeted nephrotoxic or renally cleared medications.
Pre-assignment Details: Patients who were dialyzed prior to the first serum creatinine change event or identified as a dialysis patient through a dialysis flag order, in addition to those admitted to renal transplant, liver transplant, or nephrology services were excluded.
Period: Overall Study
Arm/Group | Dashboard | Control
Started | 200 | 196
Completed | 200 | 196
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dashboard | Control | Total
Number analyzed (Participants) | 200 | 196 | 396
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 120 | 231
  >=65 years | 89 | 76 | 165
Age Continuous [Mean (Standard Deviation); unit: years] | 60.7 (16.8) | 58.3 (15.7) | 59.5 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 77 | 171
  Male | 106 | 119 | 225
Region of Enrollment [Number; unit: participants]
  United States | 200 | 196 | 396

OUTCOME MEASURES:

1. Primary Outcome: Adverse Drug Events or Potential Adverse Drug Events
Description: Our primary outcome measured the rate of AKI-related ADEs and pADEs. We defined pADEs as incidents with the potential for injury related to a drug, such as use of a non-steroidal anti-inflammatory drug for at least 24 hours, and ADEs as injuries resulting from the administration of a drug, such as a toxic vancomycin trough level or a bleed after administration of enoxaparin. We measured outcomes after completion of the inpatient encounter (either by death or discharge); pADEs or ADEs occurring after patient discharge were not included in the analysis.
Time Frame: Until patient discharge (~2 week average)
Measure: Number; unit: Patient-Medication Pairs
Units Other Than Participants: Patient-Medication Pairs
Arm/Group | Dashboard | Control
Number analyzed (Participants) | 200 | 196
Number analyzed (Patient-Medication Pairs) | 1396 | 1303
Patient-Medication Pairs | 99 | 104

2. Secondary Outcome: Time to Provider Response
Description: Time from study event to modification or discontinuation of targeted medication
Time Frame: Until patient discharge (~2 week average)
Measure: Median (Inter-Quartile Range); unit: Hours
Units Other Than Participants: Patient-Medication Pairs
Arm/Group | Dashboard | Control
Number analyzed (Participants) | 200 | 196
Number analyzed (Patient-Medication Pairs) | 1396 | 1303
Hours
  Ordered Prior to AKI | 23.7 [5.61 to 57.67] | 27.31 [5.98 to 62.57]
  Ordered After AKI | 42.37 [17.9 to 77.93] | 43.83 [17.62 to 80.58]

ADVERSE EVENTS:
Arm/Group | Dashboard | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No